CLINICAL TRIAL: NCT04835857
Title: Comparison of Cuff-Less Wrist Wearable to Cuff Based Commercial Available Blood Pressure Measuring Devices in Health Volunteers With Normal or High Blood Pressure
Brief Title: Comparison of Cuff-Less Wrist Wearable Blood Pressure Device to Cuff Based Blood Pressure Measuring Devices
Status: Recruiting | Type: Observational
Sponsor: Dynocardia, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TBPI001
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Healthy
Keywords: Blood Pressure, Cuff less, Wearable, BP
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Experimental-Arm: For the same subject,
  1. ViTrack wrist cuff is applied on one of the wrist
  2. Standard Oscillometric cuff is applied to the brachial artery / wrist of the same arm
  3. Auscultatory cuff is applied to the brachial artery of the same arm
  Interventions: Device: ViTrack; Device: Oscillometric BP Device; Device: Auscultatory cuff

INTERVENTIONS:
Device: ViTrack — ViTrack is a continuous non-invasive wearable blood pressure cuff.
Device: Oscillometric BP Device — Oscillometric blood pressure measurement is the standard of care for measuring blood pressure in outpatient / home settings.
Device: Auscultatory cuff — The auscultatory method is the gold standard for clinical blood pressure measurement. A brachial cuff is mounted and a trained healthcare provider uses a sphygmomanometer and listens for the Korotkoff sounds using a stethoscope to measure blood pressure.

SUMMARY:
(1) To compare cuff-less wrist wearable radial artery blood pressure measurements utilizing ViTrack(developed by Dynocardia) to the cuff based commercially available blood pressure device, in healthy volunteers with normal or high blood pressure.

DETAILED DESCRIPTION:
(1) The ViTrack is strapped over the radial artery at the wrist. The ViTrack blood pressure cuff will be utilized to obtain blood pressure(BP) readings in the volunteers with normal or high blood pressure. The readings from the ViTrack will be compared with the readings of a cuff-based, commercially available BP measuring device placed on the same arm.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteers 18 years and above; equal numbers of males and females to address Sex As a Biological Variable (SABV); and in sinus rhythm.
* Agree to commit to participate in the current protocol.
* Provide written informed consent prior to any study procedures being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read).

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Any other condition that would increase the risk of participation in the study in the opinion of the site Investigator.
* A difference of >10 mm Hg in left versus right arm oscillometric systolic BP.
* Upper extremity arteriovenous hemodialysis shunt.
* Wrist distortion or pain from arthritis.
* Prior trauma or surgery at the radial artery monitoring site.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of Diastolic Blood Pressure | up to 30 minutes
  3 sets readings compared across blood pressure (mmHg)
Comparison of Systolic Blood Pressure | up to 30 minutes
  3 sets readings compared across blood pressure (mmHg)

SECONDARY OUTCOMES:
Skin Irritation | Up to 72 hours
  Examining for local skin irritation

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Thanikachalam, MD, Principal Investigator — Dynocardia, Inc
Locations (1):
- Dynocardia Inc, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Personal and medical information will stay confidential and secure and will be protected in accordance with current US law. All participants will be provided with a unique ID number. All participants' information such as participants' name and address as well as background information will be de-identified to protect subject confidentiality.
  Dynocardia or its designees will comply with all relevant data collection laws when collecting data for this study. Study databases will not include the participants name or address. Images will be captured by ViTrack under patient's ID in an electronic database. All other data will be de-identified for review purpose and transferred via a secure method.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available following data analysis within 6 month of study completion and will remain available for up to 3 years.
Access Criteria: Data will be accessed via secure methods outlined in a data sharing agreement